CLINICAL TRIAL: NCT01588769
Title: A Phase I Study to Investigate Tolerability and Efficacy of Autologous Lymphoid Effector Cells Specific Against Tumour-cells (ALECSAT) Administered to Patients With Glioblastoma Multiforme (GBM)
Brief Title: A Phase I Study to Investigate Tolerability and Efficacy of ALECSAT Administered to Glioblastoma Multiforme Patients
Acronym: ALECSAT-GBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CytoVac A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV003; 2011-002180-22 (EudraCT Number)
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Brain cancer; Immunotherapy; Cell based therapy; Autologous cell based therapy; Adoptive immunotherapy; Cytotoxic T cells; Natural Killer cells
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One arm (Experimental): 3 doses of ALECSAT cell based immunotherapy planned for all enrolled patients
  Interventions: Biological: ALECSAT cell based immunotherapy

INTERVENTIONS:
Biological: ALECSAT cell based immunotherapy — I.V. injected Cell Based Medicinal Product, containing between 10 million and one billion autologous Cytotoxic T cells and Natural Killer cells.

SUMMARY:
It is the primary objective of this study to show safety and tolerability for administration of the cell based immunotherapy ALECSAT to patients with Glioblastoma brain cancer. It is a secondary objective to establish if any indications of positive therapeutic or palliative effects may be observed.

DETAILED DESCRIPTION:
The primary objective for this study is to establish if any side effects or toxicity issues occur, that will prevent further clinical development of the autologous cell based immunotherapy ALECSAT in Glioblastoma (GBM) or to establish if there are side effects or toxicity issues, that will suggest that the further clinical development planned, has to change course significantly. It is a primary objective to show safety and tolerability for administration of ALECSAT, thus not meeting this endpoint, may stop further clinical development of ALECSAT.

The secondary objective for this study is to establish if any indications of a positive therapeutic or palliative effect may be observed. As this is a secondary objective, no observed significant positive clinical effect, will not prevent further clinical development or in itself, trigger changes in the further clinical development planned.

The overall endpoint of the study is to develop a new therapeutic approach that may slow down or stop disease progression in late stage GBM patients.

ALECSAT is an autologous cell based immunotherapy based on the patient's own Natural Killer cells and CytoToxic T cells. The cells are isolated from the patient's own blood - activated and expanded in number before re administering i. v.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrence of GBM tumour documented by MRI and PET in patients having received all available standard treatment.
2. Be over the age of 18 and capable of understanding the information and giving informed consent.
3. Adequate performance status > 50% (see below*).

   * Performance is monitored according to the Karnofsky Performance Score (KPS)

     * 100% - normal, no complaints, no signs of disease
     * 90% - capable of normal activity, few symptoms or signs of disease
     * 80% - normal activity with some difficulty, some symptoms or signs
     * 70% - caring for self, not capable of normal activity or work
     * 60% - requiring some help, can take care of most personal requirements
     * 50% - requires help often, requires frequent medical care
     * 40% - disabled, requires special care and help
     * 30% - severely disabled, hospital admission indicated but no risk of death
     * 20% - very ill, urgently requiring admission, requires supportive measures or treatment
     * 10% - moribund, rapidly progressive fatal disease processes
     * 0% - death.

Exclusion Criteria:

1. A low blood count (haemoglobin < 6.0 mmol/l).
2. Lymphocyte counts below 0.8 x 109/l.
3. Positive tests for anti-HIV-1/2;
4. Positive tests for HBsAg,
5. Positive tests for anti-HBc and Anti-HCV.
6. Syphilis i.e. being positive in a Treponema Pallidum test.
7. Uncontrolled serious bacterial, viral, fungal or parasitic infection.
8. Clinically significant autoimmune disorders or conditions of immune suppression.
9. Treatment with chemotherapy three weeks prior to inclusion in the clinical trial.
10. Pregnant women cannot be included in the trial. Fertile women can only be included with a negative pregnancy test and must use contraceptives during the study.
11. Blood transfusions within 48 hours prior to donation of blood for ALECSAT production.
12. Inclusion in other clinical trials 6 weeks prior to inclusion in the trial.
13. The patient's medical condition is evaluated to be so poor that there is a significant risk for the patient to be part of the trial and to evaluate any effects of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Observation of tolerability and sideeffects of treatment monitored by objective medical examinations, Karnofsky score and QOL interviews. | 3 months

SECONDARY OUTCOMES:
Potential clinical effect will be monitored by PET-MRI and SPECT scanning of the brain. | 3 months
  A total of 4 scanannings are performed during the study: 2 PET-MRI scans and 2 SPECT (Single-photon emission computed tomography) scans.

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Jensen, PhD, Study Director — CytoVac A/S (Sponsor)
Locations (1):
- Department of Neurosurgery, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided